CLINICAL TRIAL: NCT00002705
Title: TOPOTECAN FOR CHILDREN WITH REFRACTORY LEUKEMIA, A PEDIATRIC ONCOLOGY GROUP PHASE I COOPERATIVE AGREEMENT STUDY
Brief Title: Topotecan in Treating Children With Refractory Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01833; POG-9575; CDR0000064511 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2001-05

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Topotecan

ARMS (1):
- Arm I (Experimental): Single-Agent Chemotherapy. Topotecan, TOPO, NSC-609699.
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
Phase I trial to study the effectiveness of topotecan in treating children with refractory leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Describe the qualitative and quantitative toxic effects, including acute and chronic dose-limiting toxicity, cumulative toxicity, and time to recovery, in pediatric patients with refractory leukemia who are treated with a 30-minute daily infusion of topotecan (TOPO) for up to 12 consecutive days every 3 weeks.

II. Estimate the maximum tolerated dose of TOPO that results in tolerable, predictable, and reversible toxicity.

III. Determine the precautions and supportive therapy that should be used and the clinical and laboratory studies needed to monitor or alter therapy to prevent unacceptable toxicity in these patients.

IV. Observe any antileukemic effects that may occur during this phase I study in which duration of treatment is increased from 7 to 9 and then 12 days and TOPO doses are escalated.

V. Determine the recommended phase II pediatric dose of TOPO. VI. Characterize the pharmacokinetic parameters of TOPO and evaluate changes in these parameters with the first and last doses to determine whether there is drug accumulation.

VII. Correlate, if possible, these pharmacokinetic parameters with clinical response and toxicity.

OUTLINE:

Single-Agent Chemotherapy. Topotecan, TOPO, NSC-609699.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

-Histologically or cytologically confirmed leukemia refractory to conventional therapy or for which no effective curative therapy exists

PATIENT CHARACTERISTICS:

* Age: Under 21
* Performance status: ECOG 0-2
* Life expectancy: At least 8 weeks
* Adequate platelet count and hemoglobin required (transfusion allowed)
* Bilirubin no greater than 1.5 mg/dL
* AST or ALT no greater than 2 times normal
* Creatinine less than 1.5 mg/dL
* Adequate nutritional status, e.g. higher than third percentile weight for height
* Albumin at least 3 g/dL
* No severe uncontrolled infection
* No pregnant women
* Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since systemic chemotherapy (6 weeks since nitrosoureas)
* Recovered at least 3 months since bone marrow transplant (at least 6 months since total-body irradiation)
* No concurrent anticancer therapy
* No concurrent treatment studies

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 1996-04; Primary Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Lee Furman, MD, Study Chair — St. Jude Children's Research Hospital
Locations (31):
- United States (27):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Memorial Mission Hospital, Asheville, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland

REFERENCES:
- [Result] Furman WL, Stewart CF, Kirstein M, Kepner JL, Bernstein ML, Kung F, Vietti TJ, Steuber CP, Becton DL, Baruchel S, Pratt C. Protracted intermittent schedule of topotecan in children with refractory acute leukemia: a pediatric oncology group study. J Clin Oncol. 2002 Mar 15;20(6):1617-24. doi: 10.1200/JCO.2002.20.6.1617. PMID 11896112